CLINICAL TRIAL: NCT02469896
Title: A Phase 2 Randomized, Placebo Controlled Trial of Tocilizumab in ALS Subjects
Brief Title: A Trial of Tocilizumab in ALS Subjects
Acronym: TCZALS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barrow Neurological Institute (Other)
Collaborators: ALS Association (Other); Barrow Neurological Foundation (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Shafeeq Ladha, MD, Director, Gregory W. Fulton ALS and Neuromuscular Disease Center, Barrow Neurological Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015TCZALS-001
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease; Motor Neuron Disease
Keywords: ALS; tocilizumab; biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 8 subjects will receive matching IV placebo every 4 weeks for 3 months.
  Interventions: Other: Placebo
- Active drug (Active Comparator): 14 subjects will receive 8mg/kg of IV tocilizumab every 4 weeks for 3 months.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — IV Infusion
  Other Names: Actemra
  Arms: Active drug
Other: Placebo — IV Infusion
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This research study is being done to find out if tocilizumab, also known as Actemra™, can help with Amyotrophic Lateral Sclerosis (ALS). The investigators also want to find out if tocilizumab is safe to take without causing too many side effects.

Currently ALS has no cure and 2 modestly effective treatment to slow the progression of the disease. Although not the initial cause of ALS, the immune system plays a role in the death of motor neurons. The immune cells that participate in this process are stimulated by a substance called interleukin-6 (IL-6) whose effect is blocked by tocilizumab and thus, may slow the death of motor neurons and slow the disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled 16-week study evaluating the safety and tolerability of tocilizumab in subjects with ALS.

The primary objective of the study is to determine the safety and tolerability of intravenous administration of 8 mg/kg of tocilizumab every 4 weeks vs. matched intravenous placebo administered every 4 weeks over an 8 week period.

The secondary objectives of the study are to describe the expression of pro-inflammatory genes in Peripheral Blood Mononuclear Cells (PBMCs) of sporadic ALS patients, to assess the ability of tocilizumab to reduce the expression of pro-inflammatory genes in PBMCs and pro-inflammatory cytokines in the cerebrospinal fluid (CSF) of patients with sporadic ALS and to assess the CSF penetration of tocilizumab. Mean peripheral benzodiazepine receptor 28 (PBR28) uptake will be measured in the motor cortices as regions of interest (ROIs), and will be compared between pre- and post-dose, for Massachusetts General Hospital (MGH) subjects.

Approximately 5 Northeast ALS Consortium (NEALS) Centers in the US will participate in the study. Twenty-four subjects will be randomized in the study.

This study will be conducted in subjects who meet the El Escorial criteria of possible, laboratory-supported probable, probable, or definite criteria for a diagnosis of ALS. At screening, eligible subjects must be at least 18 years old, must have a slow vital capacity (SVC) ≥ 40% of predicted capacity for age, height and gender (and in the opinion of the investigator is able to comply with and complete the trial), and must provide written informed consent prior to screening. Subjects on a stable dose of riluzole and those not taking riluzole, and women of child-bearing age at screening are eligible for inclusion as long as they meet specific protocol requirements. Detailed criteria are described in the body of the protocol.

Subjects participating in the magnetic resonance imaging - positron emission tomography (MRI-PET) portion of the study (MGH only) must meet the following additional criteria.High or mixed affinity to bind translocator protein (TSPO) (Ala/Ala or Ala/Thr,) Upper Motor Neuron Burden (UMNB) Scale Score ≥25 (out of 45) at the Screening Visit.

and have the ability to safely undergo MRI-PET scans based on the opinion of the site investigator.

Subjects will be randomly assigned in a 2:1 ratio to intravenous tocilizumab 8 mg/kg or matching placebo every 4 weeks over an 8 week period.

This research study protocol allows the subject to receive up to 3 infusions of Tocilizumab. Even if the treatment is shown to be of benefit, additional infusions of Tocilizumab beyond that allowed in the protocol cannot be given to the subject while she/he is participating in this study.

Subjects will remain on randomized, placebo-controlled, double-blind treatment until the Week 8 visit. Each randomized subject will also have a Week 12 Follow-up visit and Week 16 End-of-Study visit to assess for adverse events (AEs), changes in concomitant medications, to administer the ALS Functional Rating Scale (ALSFRS-R) and selected study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ALS (El Escorial criteria: possible, laboratory-supported probable, probable or definite)
* Capable of providing informed consent and complying with trial procedures.
* High inflammatory profile of PBMC gene expression
* Upright SVC ≥40% of predicted value for gender, height and age at Screening and in the opinion of the investigator is able to comply with and complete the trial.
* Women must not be able to become pregnant for the duration of the study.
* Negative tuberculosis blood or skin test at Screening
* Not taking riluzole, or on a stable dosage for at least 30 days prior to Screening.
* Subjects medically able to undergo lumbar puncture (LP)
* Subjects must agree not to take live attenuated vaccines 30 days before Screening, throughout the duration of the trial and for 60 days following the subject's last dose of study drug
* Geographic accessibility to the study site

Additional MRI-PET Inclusion Criteria (MGH only):

* High or mixed affinity to bind TSPO protein (Ala/Ala or Ala/Thr) (see section 7.1)
* Upper Motor Neuron Burden (UMNB) Scale Score ≥25 (out of 45) at the Screening Visit.
* Able to safely undergo MRI-PET scans based on the opinion of the site investigator.

Exclusion Criteria:

* Prior use of Tocilizumab, cell-depleting therapies, alkylating agents, total lymphoid irradiation
* Stem cell therapies
* Dependence on mechanical ventilation as defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use
* Presence of tracheostomy at Screening
* Exposure to any anti-inflammatory agent currently under investigation for the treatment of patients with ALS (off label use or investigational) within 30 days prior to the Screening Visit (examples include NP001 and Lunasin). Medications that do not have an anti-inflammatory mechanism, such as mexiletine or retigabine are allowed if on stable dose for 30 days prior to Screening visit
* Treatment with a prohibited medication within 30 days of the Screening Visit
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of Screening
* Presence of diaphragm pacing system at Screening.
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation
* History of or active diverticulitis, diverticulosis requiring antibiotic treatment, peptic ulcer disease, or gastrointestinal (GI) tract perforation, or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis or other symptomatic lower GI conditions that might predispose to perforations
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections.
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Presence of any of the following clinical conditions: bleeding diathesis, or any other clinical condition that would, in the opinion of the investigator, place the patient at increased risk during LP. Drug abuse or alcoholism within the past 12 months. Unstable cardiac, pulmonary, renal, hepatic, endocrine, hematologic, or active infectious disease, including current or prior malignancy. Rheumatic autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis. Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years. Human immunodeficiency virus infection or other immunodeficient state.Uncontrolled hypertension defined as systolic blood pressure > 170 or diastolic blood pressure > 110. Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the Screening Visit
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening
* Screening alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin > than 1.5 times the upper limit of normal (ULN), serum creatinine > 1.6 mg/dL in female patients and > 1.9 mg/dL in male patients (patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rate (GFR) are >30), hemoglobin < 85 g/L, white blood cells < 3.0 x 109/L, absolute neutrophil count of <2000/mm3, absolute lymphocyte count < 0.5 x 109/L, platelet concentration of <100,000/mm3, positive Hepatitis B surface antigen (HBsAg)
* Pregnant women or women currently breastfeeding
* No history of chicken pox infection or no history of varicella zoster vaccination
* Any reason in the opinion of the investigator that the patient may not be able to comply with study procedures, complete the study or is unsuitable for immunosuppressive therapy.

Additional MR-PET Exclusion Criteria (MGH only):

* Any contraindication to undergo MRI studies such as

  * History of a cardiac pacemaker or pacemaker wires
  * Metallic particles in the body
  * Vascular clips in the head
  * Prosthetic heart valves
  * Claustrophobia
* Radiation exposure that exceeds the site's current guidelines
* Current use of tobacco products including cigarettes, e-cigarettes, cigars, snuff and chewing tobacco, or nicotine replacement products such as gum, or patch
* Taking any other anti-inflammatory or immune modulating medications except for over the counter NSAIDs
* Unwilling or unable to discontinue benzodiazepine usage (other than Lorazepam, Clonazepam, or Zolpidem) for one day prior to scanning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shafeeq Ladha, MD, Principal Investigator — Barrow Neurological Institute
Locations (5):
- United States (5):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Penn State College of Medicine Milton S. Hershey Medical Center, Hershey, Pennsylvania

REFERENCES:
- [Derived] Milligan C, Atassi N, Babu S, Barohn RJ, Caress JB, Cudkowicz ME, Evora A, Hawkins GA, Wosiski-Kuhn M, Macklin EA, Shefner JM, Simmons Z, Bowser RP, Ladha SS. Tocilizumab is safe and tolerable and reduces C-reactive protein concentrations in the plasma and cerebrospinal fluid of ALS patients. Muscle Nerve. 2021 Sep;64(3):309-320. doi: 10.1002/mus.27339. Epub 2021 Jun 24. PMID 34075589

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Drug: 16 subjects will receive 8mg/kg of IV tocilizumab every 4 weeks for 3 months.
  Tocilizumab: IV Infusion
Period: Overall Study
Arm/Group | Placebo | Active Drug
Started | 8 | 14
Completed | 6 | 14
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Drug | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (8.6) | 61.9 (8.7) | 60.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 14 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Tolerant to Study Drug
Description: Tolerability will be assessed by on the proportion of participants remaining on study drug through all 3 doses and remaining on study and free from possibly drug-related and dose-limiting SAEs to the end of follow-up. Safety will be assessed by the occurrence of severe adverse events (SAEs), overall rates of adverse events (AEs), clinically significant abnormal laboratory tests, and changes in vital signs.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Tolerability: 8 subjects will receive matching IV placebo every 4 weeks for 3 months.
  Placebo: IV Infusion
- Active Drug Tolerability: 14 subjects will receive 8mg/kg of IV tocilizumab every 4 weeks for 3 months.
  Tocilizumab: IV Infusion
Arm/Group | Placebo Tolerability | Active Drug Tolerability
Number analyzed (Participants) | 8 | 14
Participants | 6 | 12
Statistical Analysis 1: Comparison: Placebo Tolerability vs Active Drug Tolerability; Test type: Superiority; p = 0.602, Fisher Exact; Risk Ratio (RR) = 0.875, 95% CI 2-sided [0.556 to 1.377]

2. Primary Outcome: Rates of All-cause Mortality
Description: Safety will be assessed by the occurrence of all-cause mortality.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Participants
  Died | 0 | 0
  Alive | 8 | 14
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; No statistical data was obtain because no patients died during the trial

3. Secondary Outcome: Rate of Decline in Slow Vital Capacity (SVC)
Description: Efficacy will be assessed by the change in the rate of change of SVC as measured by change in percent predicted per month. The SVC is a measure of lung capacity that is reported as the percent of the predicted value expected based on gender and height. In ALS patients, this measure declines over time as a result of progressive respiratory muscle weakness.
Time Frame: 16 weeks
Population: Discrepancies in the number of subjects analyzed are a result of subjects with missed data collection during the specific time points.
Measure: Least Squares Mean (Standard Error); unit: Percentage points change per month
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Percentage points change per month | -0.765 (0.829) | -0.666 (0.560)
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.922, Mixed Models Analysis — Unadjusted; Slope = 0.099, 95% CI 2-sided [-1.902 to 2.099]

4. Secondary Outcome: Rate of Decline ALS Functional Rating Scale Revised (ALSFRS-R)
Description: Efficacy will be assessed by the mean change in ALSFRS-R total score.The ALSFRS-R scale measures the functional capabilities of an ALS patient in multiple domains such as swallowing, speech, fine motor, and breathing functions. It ranges from a maximum score of 48 for normal functioning to 0 for death or dependance on mechanical ventilation and declines by approximately 1 point per month on average for an ALS patient.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
units on a scale | -0.583 (0.313) | -0.591 (0.211)
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.983, Mixed Models Analysis; Difference of slopes = -0.008, 95% CI 2-sided [-0.761 to 0.745]

5. Secondary Outcome: Rate of Decline Handheld Dynamometry (HHD)
Description: Efficacy will be assessed by the change in the rate of change of HHD upper and lower extremity mega-scores. HHD utilizes an electronic pressure sensor to measure strength of individual muscles in kilograms. To calculate megascores, the mean and standard deviation of each muscle or muscle group, without regard to laterality, will be calculated from the baseline assessment of all participants. Strength estimates of each bilateral muscle or muscle group will be converted to Z scores by subtracting the relevant mean and dividing by the relevant standard deviation. Z scores for all upper extremity measurements (shoulder flexion, elbow flexion, elbow extension, wrist extension, and first dorsal interosseous contraction) and all lower extremity measurements (hip flexion, knee flexion, knee extension, and ankle dorsiflexion) will be averaged to yield upper and lower extremity megascores. Larger values indicate greater strength.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Z-score
  HHD Upper extremity mega-score | -0.028 (0.035) | -0.070 (0.024)
  HHD Lower extremity mega-score: number analyzed (Participants) | 7 | 14
  HHD Lower extremity mega-score | -0.018 (0.039) | -0.032 (0.026)

6. Secondary Outcome: Change in Peripheral Blood Mononuclear Cell (PBMC) Gene Expression
Description: Target engagement will be assessed by comparing the PBMC fold change in cytokine gene expression from baseline to week 4-16 average of ALS patients receiving drug versus placebo.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change in gene expression
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Fold change in gene expression
  PBMC IL-6 fold-change | 1.21 [0.60 to 2.54] | 1.39 [0.52 to 5.00]
  PBMC IL-8 fold-change | 1.33 [0.08 to 39.4] | 1.79 [0.38 to 14.8]
  PBMC Matrix Metalloproteinase 1 (MMP1)fold-change: number analyzed (Participants) | 8 | 13
  PBMC Matrix Metalloproteinase 1 (MMP1)fold-change | 1.01 [0.37 to 2.13] | 1.21 [0.42 to 3.28]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; PBMC IL-6 fold-change; Test type: Superiority; p = 0.684, t-test, 2 sided; Ratio of geometric means = 1.150, 95% CI 2-sided [0.566 to 2.337]
Statistical Analysis 2: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.663, t-test, 2 sided; Ratio of geometric means = 1.344, 95% CI 2-sided [0.331 to 2.080]
Statistical Analysis 3: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.500, t-test, 2 sided; Ratio of geometric means = 1.198, 95% CI 2-sided [0.691 to 2.080]

7. Secondary Outcome: Changes in Cytokine Levels in the Plasma
Description: Target engagement will be assessed by mean change in plasma cytokine concentration between weeks 4 and 16 in ALS subjects receiving placebo or active drug.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Fold change in concentration
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Fold change in concentration
  CRP (ug/mL): number analyzed (Participants) | 8 | 13
  CRP (ug/mL) | 1.051 [0.279 to 3.952] | 0.049 [0.019 to 0.126]
  IL-1beta (pg/mL) | 0.969 [0.608 to 1.545] | 1.266 [0.871 to 1.840]
  IL-6 (pg/mL) | 0.897 [0.532 to 1.515] | 17.974 [12.900 to 25.043]
  IL-8 (pg/mL) | 1.241 [0.862 to 1.787] | 1.569 [1.169 to 2.105]
  IL-17 (pg/mL): number analyzed (Participants) | 6 | 14
  IL-17 (pg/mL) | 0.962 [0.470 to 1.967] | 1.342 [0.809 to 2.226]
  Tumor necrosis factor (TNF)-alpha (pg/mL) | 1.180 [0.981 to 1.419] | 1.054 [0.923 to 1.204]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of fold change = 0.047, 95% CI 2-sided [0.010 to 0.217]
Statistical Analysis 2: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.247, Mixed Models Analysis; Ratio of fold change = 1.306, 95% CI 2-sided [0.828 to 2.059]
Statistical Analysis 3: Comparison: Placebo vs Active Drug; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of fold change = 19.591, 95% CI 2-sided [11.143 to 34.446]
Statistical Analysis 4: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.185, Mixed Models Analysis; Ratio of fold change = 1.264, 95% CI 2-sided [0.892 to 1.791]
Statistical Analysis 5: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.427, Mixed Models Analysis; Ratio of fold change = 1.396, 95% CI 2-sided [0.608 to 3.206]
Statistical Analysis 6: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.285, Mixed Models Analysis; Ratio of fold change = 0.893, 95% CI 2-sided [0.725 to 1.100]

8. Secondary Outcome: Change in Mean Concentration Cytokines in the Cerebrospinal Fluid (CSF)
Description: Target engagement will be assessed by the mean change in CSF cytokine concentration between baseline and week 8 in ALS subjects receiving placebo or active drug.
Time Frame: 8 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Fold change in concentration
Groups:
- Active Drug: 14subjects will receive 8mg/kg of IV tocilizumab every 4 weeks for 3 months.
  Tocilizumab: IV Infusion
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
Fold change in concentration
  CRP (ng/mL) | 0.641 [0.216 to 1.903] | 0.107 [0.044 to 0.260]
  IL-1beta (pg/mL) | 1.498 [0.542 to 4.138] | 1.110 [0.459 to 2.679]
  IL-6 (pg/mL) | 1.242 [0.781 to 1.974] | 4.115 [2.813 to 6.018]
  IL-8 (pg/mL) | 0.946 [0.758 to 1.181] | 1.020 [0.854 to 1.218]
  TNF-alpha (pg/mL) | 0.989 [0.727 to 1.346] | 1.066 [0.833 to 1.365]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.011, Mixed Models Analysis; Ratio of fold change = 0.167, 95% CI 2-sided [0.043 to 0.643]
Statistical Analysis 2: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.604, Mixed Models Analysis; Ratio of fold change = 0.741, 95% CI 2-sided [0.228 to 2.405]
Statistical Analysis 3: Comparison: Placebo vs Active Drug; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of fold change = 2.940, 95% CI 2-sided [1.823 to 4.740]
Statistical Analysis 4: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.587, Mixed Models Analysis; Ratio of fold change = 1.078, 95% CI 2-sided [0.813 to 1.431]
Statistical Analysis 5: Comparison: Placebo vs Active Drug; Test type: Superiority; p = 0.697, Mixed Models Analysis; Ratio of fold change = 1.078, 95% CI 2-sided [0.728 to 1.595]

9. Secondary Outcome: Change in CSF Soluble Interleukin-6 (sIL-6) Receptor Concentrations
Description: Target engagement will be assessed by comparing the mean change in CSF sIL-6 receptor concentrations (ng/mL) between baseline and week 8 of the placebo and active drug groups.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 8 | 14
ng/mL | 1.029 [0.886 to 1.195] | 1.836 [1.621 to 2.080]
Statistical Analysis 1: Comparison: Placebo vs Active Drug; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of fold change = 1.785, 95% CI 2-sided [1.502 to 2.121]

10. Secondary Outcome: Peripheral Benzodiazepine Receptor 28 (PBR28) Positron Emission Tomography (PET)
Description: Measure the effects of tocilizumab on reducing glial activation measured by PBR28 PET in a subset of trial participants.
Time Frame: 8 weeks
Population: Only 2 patients met inclusion criteria for the PET portion of the study and thus, the data could not be statistically analyzed.
Measure: Number; unit: Standardized Uptake Variable Ratio(SUVR)
Arm/Group | Placebo | Active Drug
Number analyzed (Participants) | 1 | 1
Standardized Uptake Variable Ratio(SUVR)
  Baseline | 1.225282 | 1.059685
  Week 8 | 1.361542 | 1.056888

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study lasting up to 16 weeks in each subject.
Arm/Group | Placebo | Active Drug
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/14
Other Adverse Events (participants affected / at risk) | 6/8 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Active Drug (N=14)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Active Drug (N=14)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear Pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Catheter Site Related Reaction (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 2 (2)
Infusion Site Pruritus (General disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 1 (1)
Puncture Site Pain (General disorders) | 4 (4) | 2 (2)
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Gingival Abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 3 (4)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (2) | 3 (4)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 2 (2)
Platelet Count Increased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02469896/Prot_SAP_000.pdf